CLINICAL TRIAL: NCT06996847
Title: Effectiveness of a Psychoeducational Program to Promote a Critical Attitude Towards the Symbolic Consumption of Yoghurt in Primary School Children: Randomized Clinical Trial
Brief Title: A Protocol to Promote Critical Consumption (PCC)
Acronym: PCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de San Martín de Porres (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001-2025-IDI-FCCTP
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Promote a Critical Attitude Towards the Symbolic Consumption of Youghurt in Primary School Children
Keywords: Child Behavior; Intervention / Treatment; Mental Health/education; Psychosocial Functioning; Feeding Behavior
MeSH Terms: conditions — Child Behavior; Psychological Well-Being; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): The promotion of critical consumption in children is to be developed in primary school classrooms. Students will spend a total of 7 hours: (2 sessions of 1 hour per week) for 3 consecutive weeks, plus a feedback session (1 hour per week); and there will be another session with parents (1 hour per week). The psychologist tutor will receive a set of six activities related to discriminating between symbolic and critical yoghurt consumption in children, understanding the persuasive intent of yoghurt advertising, awareness of social pressure and critical attitude. Psychological tutors will be trained and provided with support materials and equipment.
  Interventions: Behavioral: psychoeducational programme to promote a critical attitude towards the symbolic consumption of yoghurt in primary school children
- Protocol to encourage critical consumption (Other): As detailed in the description for the intervention group, the psychologist tutors guide the students in the classroom for two hours per week for three weeks in a row, plus a feedback session. There will also be a session with parents.
  Interventions: Behavioral: psychoeducational programme to promote a critical attitude towards the symbolic consumption of yoghurt in primary school children
- No Intervention: Control (No Intervention): Five months after the start of the randomised clinical trial, primary school teachers in the control group will receive an unguided version of the psychoeducational intervention programme, supplemented by an online peer support group. They will be provided with the six activities related to critical consumption and awareness of the persuasive intent of advertising and social pressure for students to practice independently, in addition to online support from the research group. As in the intervention group, psychological support will be provided to children with emotional difficulties.

INTERVENTIONS:
Behavioral: psychoeducational programme to promote a critical attitude towards the symbolic consumption of yoghurt in primary school children — The promotion of critical consumption in children is to be developed in primary school classrooms. Students will spend a total of 7 hours: (2 sessions of 1 hour per week) for 3 consecutive weeks, plus a feedback session (1 hour per week); and there will be another session with parents (1 hour per week). The psychologist tutor will receive a set of six activities related to discriminating between symbolic and critical yoghurt consumption in children, understanding the persuasive intent of yoghurt advertising, awareness of social pressure and critical attitude. Psychological tutors will be trained and provided with support materials and equipment
  Arms: Intervention group; Protocol to encourage critical consumption

SUMMARY:
The aim of this randomised controlled trial is to evaluate the efficacy of an intervention called a psychoeducational programme to promote a critical attitude towards the symbolic consumption of yoghurt in primary school children. Specifically, a cluster randomised controlled trial will be conducted in primary schools in Lima, Peru. After informed consent of the tutor psychologists, children and parents, schools will be randomly assigned, in a 1:1 ratio, to the intervention or control group, with a total of 240 fourth grade students and 24 tutor psychologists. The primary and secondary research questions are as follows.

DETAILED DESCRIPTION:
The aim of this randomised controlled trial is to evaluate the efficacy of an intervention called a psychoeducational programme to promote a critical attitude towards the symbolic consumption of yoghurt in primary school children.

Specifically, a cluster randomised controlled trial will be conducted in primary schools in Lima, Peru. After informed consent of the tutor psychologists, children and parents, schools will be randomly assigned, in a 1:1 ratio, to the intervention or control group, with a total of 240 fourth grade students and 24 tutor psychologists. The primary and secondary research questions are as follows.

The primary research question:

• Is the intervention effective in fostering critical attitudes towards symbolic yoghurt consumption in children from pre-test to post-test (Record of symbolic consumption responses: self, parent and facilitator reports)?

The secondary research questions:

* Is the intervention effective in stabilising the child's deductive skills?
* Is the main question moderated by the child's gender, physical disability, dysfunctional state and the facilitator's experience? The intervention will take place in the school classroom (2 sessions of 1 hour per week) for 3 consecutive weeks, plus a feedback session (1 hour per week); and a further session with parents (1 hour per week). A set of participatory techniques will be included to help distinguish between symbolic and nutritional aspects of yoghurt (e.g. role play), to help understand the persuasive intent of advertising (e.g. opinion wheel), and to help balance between peer pressure consumption and critical attitude. The control group will carry out the usual teaching and will receive the set of activities after the end of the trial. After two interviews with the child and another interview with the parents, the Symbolic Consumption Response Register will be completed, and the Raven's Progressive Matrices Test-2 will be applied before and immediately after the intervention, both in the control group and in the intervention group. The facilitators of both groups will complete a form immediately after the end of each psychoeducational activity for both children and parents Eligibility Criteria Description Additional inclusion criteria for schools are: (a) access to the classroom within the school, and (b) written informed consent for participation in this study by the 4th grade primary school psychologists. Inclusion criteria for children are: (a) enrolled in 4th grade, (b) give informed consent, (c) have written informed consent from their parents or legal guardians, present normal intelligence according to the Raven's Progressive Matrices Test-2.

ELIGIBILITY:
Inclusion Criteria:

For children:

* Enrolled in 4th grade
* Provide informed assent
* Have written informed consent from their parents or legal guardians
* Present normal intelligence according to the Raven's Progressive Matrices Test-2

For schools:

* Provide access to the classroom within the school
* Provide written informed consent for participation from 4th grade primary school psychologists

Exclusion Criteria:

* Not enrolled in 4th grade
* Suffering from a mental disorder
* Repeating 4th grade
* Below normal intelligence according to the Raven-2 Progressive Matrices Test

Ages: 9 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Change from the child's initial symbolic consumption at 6 weeks | Baseline, 6 weeks
  The Symbolic Consumption Response Register (CRR) consists of 15 questions that are used to assess children's attitudes related to symbolic consumption. The frequency of children's symbolic consumption responses during the past week is rated on a 17-point scale (lowest frequency of symbolism = 1-4; intermediate frequency of symbolism = 5-13; highest frequency of symbolism = 14-17). Responses will be examined as an overall result and separately on understanding the persuasive intent of yoghurt advertising, on awareness of peer pressure and on critical attitude to consumption. Information for recording responses will be obtained from two interviews with the child and one interview with the parents, and from the six psychoeducational strategies developed with the children and one session with the parents. The answers of the children and their parents will be reported orally. The responses will be analysed separately.
Change from the child's initial symbolic consumption at 19 weeks | Baseline, 19 weeks
  The Symbolic Consumption Response Register (CRR) consists of 15 questions that are used to assess children's attitudes related to symbolic consumption. The frequency of children's symbolic consumption responses during the past week is rated on a 17-point scale (lowest frequency of symbolism = 1-4; intermediate frequency of symbolism = 5-13; highest frequency of symbolism = 14-17). Responses will be examined as an overall result and separately on understanding the persuasive intent of yoghurt advertising, on awareness of peer pressure and on critical attitude to consumption. Information for recording responses will be obtained from two interviews with the child and one interview with the parents, and from the six psychoeducational strategies developed with the children and one session with the parents. The answers of the children and their parents will be reported orally. The responses will be analysed separately.

SECONDARY OUTCOMES:
Stability of child's deductive ability at 6 weeks | Baseline, 6 weeks
  Raven's Progressive Matrices Test-2 (RPM-2) is composed of 12 non-verbal colour items out of a total of 36, which allows the assessment of deductive ability independently of the knowledge acquired by children aged 9-12 years. The deductive ability at the time of assessment shall be determined on a 12-point scale (inadequate deductive level < 8 points; adequate deductive level = 8-12 points). The score achieved will be the expected result. The response record will be obtained from the child's non-verbal responses.
Stability of child's deductive ability at 19 weeks | Baseline, 19 weeks
  Raven's Progressive Matrices Test-2 (RPM-2) is composed of 12 non-verbal colour items out of a total of 36, which allows the assessment of deductive ability independently of the knowledge acquired by children aged 9-12 years. The deductive ability at the time of assessment shall be determined on a 12-point scale (inadequate deductive level < 8 points; adequate deductive level = 8-12 points). The score achieved will be the expected result. The response record will be obtained from the child's non-verbal responses.
Children's assessment of the psychoeducational programme | 6 weeks
  An item is inserted for the children to answer their appreciation of the development of the psychoeducational programme (1=bad; 2=average= 3=good). It will be asked in the post-test to the children in the intervention group.
Child's Sex | Baseline
  The sex of the participants (male, female) will be obtained from the psycho-pedagogical records of each school. This aspect will be considered as a moderating factor.
Assessment of facilitators' performance | Baseline
  Two questions were constructed: one to assess the quality of performance and one to assess the experience of the facilitators. Higher scores indicate excellent performance = 4-5 points; good performance = 3 points; fair performance = 2 points; poor performance = 1 point. This assessment will be considered in the moderator performance rubric.
Children's psychosocial or behavioral dysfunction | Baseline
  Children with physical disabilities or diagnosed learning disabilities (e.g. reading comprehension deficits) will be identified in the child's psycho-pedagogical records in each school. These aspects will be considered as moderating factors.

OTHER OUTCOMES:
Adherence Assessments: Facilitator's registration | Weekly during the intervention phase (6 weeks) in the intervention group
  The facilitators of the psychoeducational program will use a form to record the events scheduled for each psychoeducational activity for both the children and their parents. The name, date, and duration of the activity will be documented. Records will be kept on each of the 5 participatory techniques, the story, the exhibition of 2 advertising videos on YouTube and the exhibition of 10 advertising posters. This information will be used to evaluate the quality of implementation of the interventions. To accomplish the full implementation of the psychoeducational programme, a total of 8 hours of intervention (2 sessions of 1 hour each per week) for 3 consecutive weeks and a 1 hour feedback session plus a 1 hour session with the parents are required. To stimulate a critical attitude towards symbolic consumption, a total of 8 psychoeducational activities should be carried out. In addition, the scores resolved in the 'B' series of the Raven's Progressive Matrices Test-2 (deductive capacity)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fidel Abregú Tueros, PhD, Principal Investigator — Research Institute, FCCTP, San Martin de Porres University, Peru

IPD SHARING:
Plan to Share IPD: Undecided
It will be subject to the authorization of the children's parents and guardians

REFERENCES:
- [Background] Money R, Wilde S, Dawson D. Review: The effectiveness of Theraplay for children under 12 - a systematic literature review. Child Adolesc Ment Health. 2021 Sep;26(3):238-251. doi: 10.1111/camh.12416. Epub 2020 Aug 6. PMID 32767491
- [Background] Lebiger-Vogel J, Rickmeyer C, Leuzinger-Bohleber M, Meurs P. Fostering Emotional Availability in Mother-Child-Dyads With an Immigrant Background: A Randomized-Controlled-Trial on the Effects of the Early Prevention Program First Steps. Front Psychol. 2022 Apr 7;13:790244. doi: 10.3389/fpsyg.2022.790244. eCollection 2022. PMID 35465509
- [Background] Vanderbilt KE, Andreason C. The influence of popular media characters on children's object choices. Br J Dev Psychol. 2023 Mar;41(1):1-12. doi: 10.1111/bjdp.12434. Epub 2022 Oct 12. PMID 36224492
- [Background] Triece P, Massazza A, Fuhr DC. Effectiveness and implementation outcomes for peer-delivered mental health interventions in low- and middle-income countries: a mixed-methods systematic review. Soc Psychiatry Psychiatr Epidemiol. 2022 Sep;57(9):1731-1747. doi: 10.1007/s00127-022-02294-y. Epub 2022 Apr 29. PMID 35484436
- See also: ASSOCIATED SOCIAL SYMBOLISM AND MANIPULATIVE ATTITUDES TOWARDS CHILDREN FROM THE PERUVIAN AMAZON — https://www.scielo.br/j/psoc/a/rZTCVbJpDBFbt7hkVNJvRZj/abstract/?lang=en
- See also: Guidelines on mental health promotive and preventive interventions for adolescents: helping adolescents thrive — https://www.who.int/publications/i/item/guidelines-on-mental-health-promotive-and-preventive-interventions-for-adolescents
- See also: Evolución del razonamiento analógico en niños: seguimiento desde los seis hasta los once años de edad — http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S1794-47242009000100007